CLINICAL TRIAL: NCT02867566
Title: A Multicenter, Randomized, Double-blind, Controlled, Phase III Study to Evaluate the Efficacy and Safety of IBI301 (Recombinant Chimeric Anti-CD20 Monoclonal Antibody ) in Combination With CHOP Regimen Versus Rituximab in Combination With CHOP Regimen in Treatment-naïve Patients With Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: A Study Comparing the Efficacy and Safety Between I-CHOP and R-CHOP in Untreated CD20-Positive Diffuse Large B-cell Lymphoma Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI301A301
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2016-08

CONDITIONS: Diffuse, Large B-Cell, Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IBI301 (Experimental): IBI301, 375mg/m2 iv q3w, 6 cycles(each cycle is 3 weeks)
  Interventions: Drug: IBI301 plus CHOP
- Rituximab (Active Comparator): Rituximab,375mg/m2 iv q3w, 6 cycles(each cycle is 3 weeks)
  Interventions: Drug: Rituximab plus CHOP

INTERVENTIONS:
Drug: IBI301 plus CHOP — Six cycles. IBI301: 375 mg/m2, IV, day 1 of each cycle; Cyclophosphamide: 750 mg/m2, IV, day 2 of each cycle; Doxorubicin: 50 mg/m2, IV, day 2 of each cycle; Vindesine: 4 mg, IV, day 2 of each cycle; Prednisone: 100 mg, po, day 2 to day 6 of each cycle.
  Arms: IBI301
Drug: Rituximab plus CHOP — Six cycles. Rituximab: 375 mg/m2, IV, day 1 of each cycle; Cyclophosphamide: 750 mg/m2, IV, day 2 of each cycle; Doxorubicin: 50 mg/m2, IV, day 2 of each cycle; Vindesine: 4 mg, IV, day 2 of each cycle; Prednisone: 100 mg, po, day 2 to day 6 of each cycle.
  Arms: Rituximab

SUMMARY:
The purpose of this study is to comparing the Efficacy and Safety between I-CHOP and R-CHOP in Untreated CD20-Positive Diffuse Large B-cell Lymphoma Patients.

ELIGIBILITY:
Inclusion Criteria:

* Untreated CD20-positive DLBCL confirmed by histopathology or cytology.
* 18 years to 75 years; Male or female patients.
* International Prognostic Index (IPI) score of 0 to 2.
* Signed an informed consent.
* At least one measurable lesions: for nodal tumor mass, more than 1.5 cm in the long axis and more than 1.0 cm in the short axis; for extranodal tumor mass, more than 1.0 cm in the long axis.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* More than 6 months life expectancy.

Exclusion Criteria:

* Participation in another interventional clinical trial in the past 3 months.
* Known allergic reactions against monoclonal antibody or rituximab.
* Contraindication to any component of CHOP regimen.
* Previous treatment for DLBCL, including chemotherapy, immunotherapy, partial radiotherapy for lymphoma, or surgical treatment (excluding tumor mass biopsies and surgical resection for non-lymphoma lesions), or prior use of any monoclonal antibody within 3 month.
* History of cytotoxic drugs treatment or anti-CD20 monoclonal antibody treatment for other disease (e.g., rheumatoid arthritis).
* Primary central nervous system (CNS) lymphoma, secondary CNS involvement, primary testicular lymphoma.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2016-08-22 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-12-26 (Actual)

PRIMARY OUTCOMES:
Overall response rate(ORR) | 18 weeks

SECONDARY OUTCOMES:
Complete remission(CR) | 18 weeks
Progression-free survival(PFS) | 1 year
Event-free survival(EFS) | 1 year
Overall survival(OS) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lugui Qiu, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Institute of Hematology; Chinese Academy of Medical Sciences, Tianjin, China

REFERENCES:
- [Derived] Song Y, Zhou H, Zhang H, Liu W, Shuang Y, Zhou K, Lv F, Xu H, Zhou J, Li W, Wang H, Zhang H, Huang H, Zhang Q, Xu W, Ge Z, Xiang Y, Wang S, Gao D, Yang S, Lin J, Wang L, Zou L, Zheng M, Liu J, Shao Z, Pang Y, Xia R, Chen Z, Hou M, Yao H, Feng R, Cai Z, Zhang M, Ran W, Liu L, Zeng S, Yang W, Liu P, Liang A, Zuo X, Zou Q, Ma J, Sang W, Guo Y, Zhang W, Cao Y, Li Y, Feng J, Du X, Zhang X, Zhao H, Zhou H, Yu J, Sun X, Zhu J, Qiu L. Efficacy and Safety of the Biosimilar IBI301 Plus Standard CHOP (I-CHOP) in Comparison With Rituximab Plus CHOP (R-CHOP) in Patients with Previously Untreated Diffuse Large B-Cell Lymphoma (DLBCL): A Randomized, Double-Blind, Parallel-Group, Phase 3 Trial. Adv Ther. 2021 Apr;38(4):1889-1903. doi: 10.1007/s12325-020-01603-8. Epub 2021 Mar 9. PMID 33751401